CLINICAL TRIAL: NCT05609760
Title: Effects of an Automated System of Pictograms to Facilitate Comprehension of Medical Indications: A Randomised Trial
Brief Title: Pictograms to Facilitate Comprehension of Medical Indications
Acronym: SIMAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Since the respiratory units have had to admit patients with covid sequelae or readmit former patients
Sponsor: Universidad de Concepcion (Other)
Collaborators: Universidad de Valparaiso (Other); Comisión Nacional de Investigación Científica y Tecnológica (Other Government); Servicio de Salud Talcahuano (Unknown); ILUSTRE MUNICIPALIDAD DE HUALPEN (Unknown); Dirección de Administración de Salud Municipal de Talcahuano (Unknown)
Responsible Party: Principal Investigator, Rosa Figueroa Iturrieta, Académica, Universidad de Concepcion
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FONDEFID19I10120
Record Dates: First submitted 2022-09-06; First posted 2022-11-08 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Asthma Chronic; Adherence, Medication; Primary Health Care
Keywords: Asthma Chronic; Adherence, Medication; Primary Health Care
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial of parallel groups with triple masking amongst patients with a recent diagnosis of asthma (<=15 days) in primary care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, clinical investigators, outcome assessors, analysts and sponsors will be kept unaware of treatment allocation. The masking of the participating patients will be carried out through an informative brochure on bronchial asthma delivered as part of the usual education, albeit without using pictograms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pictogram Group (Experimental): This intervention consists of using a pictogram system called SIMAP which was developed and validated in previous research.
  Participants allocated to this arm will received a pictographic depiction of their medical indications generated by an automated system. Information will include a description of inhaler functions, inhaler technique and correct aerochamber use.
  Interventions: Other: SIMAP
- Usual Care Group (Sham Comparator): These patients will receive their medical indications in the usual way, as established by the health team of the participating clinics. In addition, these patients will receive a bronchial asthma information leaflet as part of the usual education when explaining the disease. No pictograms will be included in these leaflets.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: SIMAP — Pictographic depiction of medical indications alongside standard communication of these recommendations.
  Arms: Pictogram Group
Other: Usual Care — Standard communication by medical staff of treatment indications for asthma. An informative leaflet will be delivered as well.
  Arms: Usual Care Group

SUMMARY:
SIMAP is a triple-masked randomised trial aimed at assessing whether an automated system of pictograms associated to medical indications results in better comprehension and adherence of said indications. Adult patients with a recent diagnosis of asthma will be randomised to receive a pictographic depiction of their treatments and recommended interventions or standard communication without assistance from their attending physician. Patients will be followed-up for 60 days using the Asthma Control Questionnaire (ACT). The primary endpoint of this study is the degree of asthma control as assessed by the aforementioned questionnaire. Secondary outcomes include the number of hospitalisations, emergency care unit visits and the need to increase bronchodilator therapy as per current Global Initiative for Asthma guidelines. Outcomes will be analysed under the intention-to-treat principle by a statistician unaware of treatment allocation.

DETAILED DESCRIPTION:
In this triple-masked randomised trial, adult participants with a recent diagnosis of asthma (<15 days) will be allocated to receive a pictographic depiction of their medical indications or a standard description of said indications. Eligible patients will include those between 18 and 65 years of age with a diagnosis of asthma established by standard clinical recommendations (clinical and spirometric criteria as established by Global Initiative for Asthma - GINA - guidelines) and in whom therapy including a bronchodilator and a controller medication (typically an inhaled steroid) is planned to be initiated. Patients with another cause of bronchial obstruction (such as COPD), those with cognitive or visual impairments that hampers the understanding of pictograms or those with a history of alcoholism or alcohol abuse will be excluded. Patients will be randomised using a permuted block sequence which shall be kept hidden from other investigators. Participants will be followed-up at seven, thirty and sixty-day intervals using the Asthma Control Questionnaire (ACT), which is the primary outcome of this study. Participants, clinical evaluators, analysts and sponsors will be kept unaware of treatment allocation. Secondary endpoints include the inhaler technique, the correct depiction of inhaler medication purpose, the rate of emergency care visits between groups, the rate of hospitalisations between groups and the need to increase bronchodilator therapy during scheduled visits within the trial. All analyses will be conducted using the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 65 years with a recent diagnosis of bronchial asthma (<=15 days) based on 2018 Global Initiative For Asthma (GINA) criteria.
* Diagnosis substantiated clinically and with consistent spirometry results as established by current GINA guidelines.
* Patients who are to initiate bronchodilator treatment, including at least one inhaled corticosteroid and one short-acting bronchodilator.

Exclusion Criteria:

* Patients presenting obstructive bronchial pathology other than bronchial asthma (chronic obstructive pulmonary disease, mixed states, etc.),
* Patients who have participated in the pictogram design phase (Stage 1 of the project),
* Patients with a diagnosis of dementia, diagnosis of harmful use of alcohol and other drugs according to the International Classification of Diseases (ICD-10).
* Patients with significant ophthalmologic pathology that prevents the use of pictograms.
* Patients who do not wish to participate in the project.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa L Figueroa, PhD, Study Director — Universidad de Concepcion; Carla Taramasco, PhD, Study Director — Universidad de Valparaiso
Locations (4):
- Chile (4):
  - Ilustre Municipalidad de San Antonio, San Antonio, Región de Valparaíso
  - Dirección de Administración de Hualpen, Hualpén, Región del Biobío
  - Dirección de Administración Salud de Talcahuano, Talcahuano, Región del Biobío
  - Corporación Municipal de Valparaiso, Valparaíso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddel HK, Bacharier LB, Bateman ED, Brightling CE, Brusselle GG, Buhl R, Cruz AA, Duijts L, Drazen JM, FitzGerald JM, Fleming LJ, Inoue H, Ko FW, Krishnan JA, Levy ML, Lin J, Mortimer K, Pitrez PM, Sheikh A, Yorgancioglu AA, Boulet LP. Global Initiative for Asthma Strategy 2021: Executive Summary and Rationale for Key Changes. Am J Respir Crit Care Med. 2022 Jan 1;205(1):17-35. doi: 10.1164/rccm.202109-2205PP. PMID 34658302
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Perez-Yarza EG, Castro-Rodriguez JA, Villa Asensi JR, Garde Garde J, Hidalgo Bermejo FJ; Grupo VESCASI. [Validation of a Spanish version of the Childhood Asthma Control Test (Sc-ACT) for use in Spain]. An Pediatr (Barc). 2015 Aug;83(2):94-103. doi: 10.1016/j.anpedi.2014.10.031. Epub 2014 Dec 30. Spanish. PMID 25555366
- [Background] Alvear G, Figueroa L, Hurtado G, Moyano L. Evaluación del grado de control del asma en un centro de atención primaria. Un estudio descriptivo. Rev. chil. enferm. respir. 2016; 32 (2): 68-76. Spanish.
- [Background] Barros IM, Alcantara TS, Mesquita AR, Bispo ML, Rocha CE, Moreira VP, Lyra Junior DP. Understanding of pictograms from the United States Pharmacopeia Dispensing Information (USP-DI) among elderly Brazilians. Patient Prefer Adherence. 2014 Oct 29;8:1493-501. doi: 10.2147/PPA.S65301. eCollection 2014. PMID 25378914

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was recruited on August 1, 2022, and concluded prematurely, with the last patient recruited on December 20, 2022. This process was meant to be conducted for six months and had an early termination in the fifth month. Patients were recruited from 5 out of the six participating health centers. Each patient provided written consent through the signature of the informed consent form. The principal investigator and the director of the healthcare center then signed this consent.
Groups:
- Pictogram Group: This intervention consists of using a pictogram system called SIMAP which was developed and validated in previous research.
  Participants allocated to this arm will received a pictographic decription of their medical indications generated by an automated system. Information will include a description of inhaler functions, inhaler technique and correct aerochamber use.
  SIMAP: Pictographic description of medical indications alongside standard communication of these recommendations.
Period: Overall Study
Arm/Group | Pictogram Group | Usual Care Group
Started | 10 | 12
Completed | 9 | 11
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The pictogram group initially consisted of 10 patients who signed the informed consent. However, after signing, one of the patients withdrew from the study and did not answer to the instruments. Despite being initially assigned to the pictogram group, we lack details about the baseline characteristics of this patient. As a result, this individual was not included in the total count of patients in the pictogram group for the baseline analysis.
Groups:
- Pictogram Group: This intervention consists of using a pictogram system called SIMAP which was developed and validated in previous research.
  Participants allocated to this arm will received a pictographic depiction of their medical indications generated by an automated system. Information will include a description of inhaler functions, inhaler technique and correct aerochamber use.
  SIMAP: Pictographic depiction of medical indications alongside standard communication of these recommendations.
- Total: Total of all reporting groups
Arm/Group | Pictogram Group | Usual Care Group | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [25 to 56] | 40.5 [28 to 57] | 37 [27 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Citizenship [Count of Participants; unit: Participants]
  Chilean | 7 | 10 | 17
  Colombian | 0 | 1 | 1
  Venezuelan | 2 | 1 | 3
Educational level [Count of Participants; unit: Participants]
  8 years of education | 0 | 1 | 1
  12 years of education | 4 | 6 | 10
  more than 12 years of education | 5 | 5 | 10
Marital status [Count of Participants; unit: Participants]
  single | 5 | 5 | 10
  married | 3 | 6 | 9
  divorced | 1 | 1 | 2
Median of ACT score baseline [Median (Inter-Quartile Range); unit: Median of ACT score] — The Asthma Control Test (ACT) evaluates the frequency of shortness of breath and other asthma symptoms, the use of rescue medications, the impact of asthma on daily activities, and individuals' overall assessment of their asthma control. The total score ranges from 5 (indicating poor asthma control) to 25 (indicating complete control), with higher scores reflecting better asthma control. A score above 19 suggests well-controlled asthma.
  Median of ACT score | 14 [13 to 16] | 16 [14 to 20] | 16 [13 to 18]
Charlson index score [Median (Inter-Quartile Range); unit: Median of the charlson score] — The Charlson Comorbidity Index (CCI) is a scale used for evaluating the overall burden of comorbid conditions in patients. It incorporates 17 chronic diseases, each assigned a specific weight based on its effect on mortality. The total score ranges from 0 to 37, with higher scores indicating more significant comorbidity and a higher risk of mortality. Comorbidity is classified as: 0-1 points (no comorbidity), 2 points (low comorbidity), and >3 points (high comorbidity).
  Median of the charlson score | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Disease Control at 60 Days
Description: 60 days after randomisation between groups using the Asthma Control Test (ACT). Min Score: 5 (indicating poor asthma control), Max Score 25 (indicating complete control). A score above 19 suggests well-controlled asthma.
Time Frame: 60 days
Population: We recruited 10 patients, who voluntarily signed the informed consent. One patient withdrew from the study after signing the informed consent, and we lost contact with another patient during the 30-day follow-up. Consequently, we were able to analyze 21 patients in the first control (7 days of follow-up) and 20 patients in the second and third follow-ups (30 days).
Measure: Median (Inter-Quartile Range); unit: Median of ACT score
Arm/Group | Pictogram Group | Usual Care Group
Number analyzed (Participants) | 9 | 11
Median of ACT score | 22 [18 to 22] | 21 [18 to 23]

2. Primary Outcome: Disease Control at 30 Days
Description: Asthma control achieved at 30 days after randomisation between groups using the Asthma Control Test (ACT).Min Score: 5 (indicating poor asthma control), Max Score 25 (indicating complete control). A score above 19 suggests well-controlled asthma.
Time Frame: 30 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Median of ACT score
Arm/Group | Pictogram Group | Usual Care Group
Number analyzed (Participants) | 9 | 11
Median of ACT score | 22 [18 to 23] | 23 [18 to 25]

3. Primary Outcome: Disease Control at 7 Days
Description: Asthma control achieved at 7 days after randomisation between groups using the Asthma Control Test (ACT). Min Score: 5 (indicating poor asthma control), Max Score 25 (indicating complete control). A score above 19 suggests well-controlled asthma.
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Median of ACT score
Arm/Group | Pictogram Group | Usual Care Group
Number analyzed (Participants) | 9 | 12
Median of ACT score | 19 [14 to 19] | 20 [15 to 22]

4. Secondary Outcome: Inhaler Technique
Description: Proper application of the inhaler technique.
Time Frame: 60 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pictogram Group | Usual Care Group
Number analyzed (Participants) | 9 | 11
Participants
  Shake the inhaler | 8 | 11
  Insert the inhaler chamber correctly. | 8 | 11
  Inhale inside the inhaler chamber. | 9 | 11
  Hold your breath for 10 seconds | 7 | 10
  Exhale inside the inhaler chamber. | 9 | 9

5. Secondary Outcome: Patient Adherence to Inhaler Technique Steps at 60 Days
Description: To assess patients' adherence to the correct inhaler technique, a five-step checklist was created, and a nurse evaluated each patient's inhalation technique. Then, the number of participants who correctly completed each individual step was reported.
Time Frame: 60 days
Population: We recruited 21 patients, who voluntarily signed the informed consent. One patient withdrew from the study after signing the informed consent, and we lost contact with another patient during the 30-day follow-up. Consequently, we were able to analyze 21 patients in the first control (7 days of follow-up) and 20 patients in the second and third follow-ups (30 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Pictogram Group | Usual Care Group
Number analyzed (Participants) | 9 | 11
Participants
  patient shakes the inhaler properly | 8 | 11
  The patient correctly attaches the air chamber to the inhaler | 8 | 11
  The patient inhales through the air chamber | 9 | 11
  The patient holds their breath for 10 seconds | 7 | 10
  The patient exhales into the air chamber | 9 | 9

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the day the intervention was applied until the end of the follow-up period (60 days). Patients were provided with the principal investigator's phone number to report any adverse events that occurred after the 60-day period. No adverse events were reported.
Description: No adverse events were reported.
Arm/Group | Pictogram Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/9 | 0/12

LIMITATIONS AND CAVEATS:
Unfortunately, the progression of the COVID-19 health crisis led to the suspension of this study. In response to the unprecedented circumstances, the study protocol underwent necessary amendments related to COVID-19 before resuming. The revised protocol with amendments received approval.

Due to the shift in priorities caused by the COVID-19 crisis, the flow of patients diagnosed with bronchial asthma was lower than anticipated in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT05609760/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT05609760/ICF_001.pdf